CLINICAL TRIAL: NCT07157982
Title: Living With Multimorbidity: Care Coordination and Symptom Management Program (COORDINATE)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IRB00500267
Record Dates: First submitted 2025-08-28; First posted 2025-09-05 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Multimorbidity
Keywords: Continuity of Patient Care; Hospital to Home Transition

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COORDINATE Program Intervention (Experimental): Participants receive the nurse-led COORDINATE Program, a nurse-led structured intervention focused on transitional care, including a discharge planning visit (pre-discharge and/or within 48 hours of discharge) and follow-ups at 1 week, 4 weeks, 6 weeks, and 3 months.
  Interventions: Behavioral: COORDINATE Program
- Enhanced Usual Care (Other): Participants receive enhanced usual care, including standard discharge teaching, a multimorbidity management toolkit, and follow-up check-ins.
  Interventions: Behavioral: Enhanced Usual Care

INTERVENTIONS:
Behavioral: COORDINATE Program — The COORDINATE Program is a nurse-led, multicomponent intervention designed to support older adults with multiple chronic conditions during their transition from hospital to home. The intervention is delivered over a 3-month period and includes the following components:
  1. Discharge Planning Visit: Conducted in person or via video, this session includes a needs assessment and shared decision-making conversation to identify participants' values and preferences.
  2. Question Prompt List: A tailored list of questions is provided to help participants engage more effectively with their care team.
  3. Goal Setting: Participants work with a nurse to identify short-term goals and action steps related to their health and care needs.
  4. Symptom Monitoring: Participants track symptoms weekly using a symptom checklist to support ongoing management and communication with providers.
  Other Names: Care Coordination and Symptom Management Program (COORDINATE)
  Arms: COORDINATE Program Intervention
Behavioral: Enhanced Usual Care — Participants in this arm will receive enhanced usual care, which includes standard discharge instructions, scheduled check-ins, and a resource toolkit with educational materials. The content includes guidance on symptom management, advance care planning, and available community resources. Participants will receive follow-up reminders and wellness checks but will not receive the structured, nurse-led intervention provided in the COORDINATE Program.
  Arms: Enhanced Usual Care

SUMMARY:
The goal of this clinical trial is to learn if a new care program, called the COORDINATE Program, can help older adults with two or more chronic health conditions. These individuals are being discharged from special hospital units called Intermediate Care Units (IMCUs), which care for people who are very sick but don't need intensive care.

The main questions this study wants to answer are:

1. Can the COORDINATE Program improve participants' quality of life?
2. Can the program reduce emergency visits, intensive care admissions, and rehospitalizations?

Researchers will compare the COORDINATE Program to the enhanced usual care with extra support to see if it works better. Participants will receive either the COORDINATE Program or enhanced usual care. They will also complete surveys at three different time points: before starting the intervention, at 3 months, and at 12 months.

For those in the COORDINATE Program group, a trained nurse will guide them through:

1. A needs assessment to find out what matters most to them
2. A list of helpful questions to ask their care team
3. Goal-setting to support managing their conditions
4. Tracking their symptoms and progress
5. Attend a discharge visit and have 5 follow-up phone or video calls over 3 months

Participants in both groups will be compensated for completing the surveys. The study hopes to improve how care is given to older adults with complex health needs and reduce unnecessary hospital visits.

DETAILED DESCRIPTION:
This study is a single-blind, two-arm randomized controlled trial (RCT) conducted at Johns Hopkins Health System IMCUs to pilot test the Care Coordination and Symptom Management (COORDINATE) Program, a multicomponent care coordination and symptom management program. The participants will be randomized 1:1 into either the COORDINATE intervention group or the enhanced usual care group. Follow-up assessments will occur at 3 and 12 months post-discharge.

Intervention Participants in the COORDINATE group will receive a structured, nurse-led intervention beginning after randomization and extending through 3 months post-discharge. The program consists of: Needs Assessment, Question Prompt List, Goals of Care Discussion, and Symptom Assessment and Tracking.

Enhanced Usual Care Participants in the enhanced usual care group receive enhanced usual care, which includes standard discharge teaching and follow-up planning by hospital staff. In addition, they are provided with a multimorbidity management toolkit developed during the co-design phase, covering communication strategies, care coordination, and resource access. A nurse also conducts discharge check-ins and follow-up calls, but without the structured components of the COORDINATE program.

ELIGIBILITY:
Inclusion Criteria:

1. aged 50 years and older
2. living with two or more chronic health conditions as identified by diagnosis in the electronic health record
3. medically complex patients defined as those admitted to intermediate care units
4. have a working telephone or contact method.

Exclusion Criteria:

1. cannot provide informed consent
2. non-English speakers
3. incapacitated or have documented cognitive impairment
4. are in hospice

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Health-related Quality of Life as Measured by the EuroQoL at 3 months | Baseline and 3 months post-discharge
  Health-related quality of life will be assessed using the EuroQoL, a widely used questionnaire that helps measure a person's overall health and quality of life. It asks about five key areas: 1) Mobility, 2) Self-care, 3) Usual daily activities, 4) Pain or discomfort, and 5) Anxiety or depression. It also includes a rating scale (0 to 100) where people mark their overall health, 0 means the worst health you can imagine, and 100 means the best.
Change from Baseline in Quality of Life as Measured by the EuroQoL at 12 Months | Baseline and 12 months post-discharge
  Health-related quality of life will be assessed using the EuroQoL, a widely used questionnaire that helps measure a person's overall health and quality of life. It asks about five key areas: 1) Mobility, 2) Self-care, 3) Usual daily activities, 4) Pain or discomfort, and 5) Anxiety or depression. It also includes a rating scale (0 to 100) where people mark their overall health, 0 means the worst health you can imagine, and 100 means the best.

SECONDARY OUTCOMES:
Difference in Number of Emergency Department Visits from Discharge to 3 Months Between the COORDINATE Program and Enhanced Usual Care | Immediately hospital discharge to 3 months post-discharge
  Emergency department (ED) visits will be tracked from hospital discharge through 3 months. Data will be collected from electronic health records and participant reports to evaluate differences between the COORDINATE Program and enhanced usual care.
Difference in Number of Emergency Department Visits from Discharge to 12 Months Between the COORDINATE Program and Enhanced Usual Care | Immediately hospital discharge to 12 months post-discharge
  Emergency department (ED) visits will be tracked from hospital discharge through 12 months. Data will be collected from electronic health records and participant reports to evaluate differences between the COORDINATE Program and enhanced usual care.
Difference in Number of Critical Care Admissions from Discharge to 3 Months Between the COORDINATE Program and Enhanced Usual Care | Immediately hospital discharge to 3 months post-discharge
  Critical care admissions, including ICU stays, will be measured from the time of discharge to 3 months post-discharge. This outcome will be used to assess whether the COORDINATE Program reduces the frequency of critical care admissions compared to enhanced usual care.
Difference in Number of Critical Care Admissions from Discharge to 12 Months Between the COORDINATE Program and Enhanced Usual Care | Immediately hospital discharge to 12 months post-discharge
  Critical care admissions, including ICU stays, will be measured from the time of discharge to 12 months post-discharge. This outcome will be used to assess whether the COORDINATE Program reduces the frequency of critical care admissions compared to enhanced usual care.
Difference in Number of All-Cause Rehospitalizations from Discharge to 3 Months Between the COORDINATE Program and Enhanced Usual Care | Immediately hospital discharge to 3 months post-discharge
  All-cause rehospitalizations will be recorded for each participant from discharge to 3 months. Data will be used to assess the impact of the COORDINATE Program on reducing readmission rates.
Difference in Number of All-Cause Rehospitalizations from Discharge to 12 Months Between the COORDINATE Program and Enhanced Usual Care | Immediately hospital discharge to 12 months post-discharge
  All-cause rehospitalizations will be recorded for each participant from discharge to 12 months. Data will be used to assess the impact of the COORDINATE Program on reducing readmission rates.

CONTACTS AND LOCATIONS:
Overall Officials: Binu Koirala, PhD, MGS, Principal Investigator — Johns Hopkins School of Nursing
Locations (1):
- Johns Hopkins Health System, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No